CLINICAL TRIAL: NCT06811909
Title: A Prospective, Multicenter, Randomized, Controlled Trial of Non-healing Venous Leg Ulcers Treated With Standard Care With or Without BR-AC
Brief Title: Non-healing Venous Leg Ulcers Treated With Standard Care With or Without BR-AC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioStem Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR-AC-VLU-101
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-infected Venous Leg Ulcer; Venous Leg Ulcer; Venous Insufficiency; Venous Stasis; Venous Reflux
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To reduce bias in the determination of closure, an independent blinded reviewer will review the image obtained from the wound measurement device in each case where the Investigator determines the wound has achieved closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR-AC plus Standard Care (Experimental): All subjects in the treatment group will receive sponsor-approved standard of care. Standard of care is defined as:
  * Sharp debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer followed by an alginate or foam pad to maintain a moist, warm wound bed, and
  * The UrgoK2™ dual compression system providing around 40 mmHg.
  Using an appropriate size to cover the entire wound area, BR-AC should be applied directly to the wound surface following sharp debridement. It is recommended that the product be trimmed to fit the area of the wound with sterile scissors before application.
  Interventions: Other: BR-AC
- Standard Care (Active Comparator): All subjects in the control group will receive sponsor-approved standard of care. Standard of care is defined as:
  * Sharp debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer followed by an alginate or foam pad to maintain a moist, warm wound bed, and
  * The UrgoK2™ dual compression system providing around 40 mmHg.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: BR-AC — BR-AC is an amnion layer, intermediate layer, and chorion layer placental membrane processed together with no separation of the layers. BR-AC is manufactured by BioStem Technologies, Inc. and is processed by the bioREtain method, which, briefly includes initial disinfection, processing with isotonic solutions, dehydration at 37-40°C, and electron beam sterilization.
  Arms: BR-AC plus Standard Care
Other: Standard Care — Standard Care is defined as:
  * Sharp debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer followed by an alginate or foam pad to maintain a moist, warm wound bed, and
  * The UrgoK2™ dual compression system providing around 40 mmHg.
  Arms: Standard Care

SUMMARY:
This study examines a patient population with a non-healing, non-infected venous leg ulcer (VLU) having adequate arterial perfusion with confirmed venous reflux. It is hypothesized that weekly applications of the human placental allograft BioREtain® Amnion Chorion (BR-AC) applied to a non-healing VLU will result in a higher proportion of wounds showing complete healing within 12 weeks of initiating therapy, compared to standard care alone.

This study has a crossover period, where subjects on standard care alone who do not achieve complete healing within 12 weeks of initiating therapy will be allowed to crossover to receive BR-AC over 12 additional weeks, to evaluate if their wound can achieve complete healing.

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, controlled study designed to evaluate the safety and efficacy of BR-AC plus standard of care versus standard of care only in the treatment of venous leg ulcers. The eligibility criteria for this study will allow for enrollment of subjects with a VLU in the range of 2 cm^2 to 20 cm^2 in area. A lower size of 2 cm^2 was selected to exclude subjects who are likely to heal under compression therapy alone.

During the two-week run-in period, subjects who show a reduction in wound area predictive of achieving complete wound closure within 12 weeks under standardized care alone (i.e., compression therapy) will be excluded from the study. Eliminating these subjects will improve the estimated treatment effect. The criteria for duration, ≥ 4 weeks but ≤ 52 weeks, allows for the selection of those wounds that have demonstrated chronicity but may still have the potential to achieve wound closure.

The trial design will control potential variables that may affect the outcome between the treatment group and the control group by standardizing the requirements for evaluating venous insufficiency confirmed by duplex Doppler ultrasound examining valvular or venous incompetence, debridement, and compression therapy. Weekly subject visits will help monitor compliance in wound care and compression therapy, as well as to document when wound closureis achieved. The study will implement the use of an electronic imaging and measurement device (eKare inSight®) using a standardized protocol to ensure the measuring of the wound surface area is accurate, highly reproducible, and minimally variable.

There will also be a crossover treatment phase for those patients that were relegated to SOC only. After their 12-week standard of care treatment phase and for only those subjects that did not achieve complete wound closure, will be allowed to crossover for an additional 12 weeks of treatment with the BR-AC product following the protocol and procedures set forth within this document.

A follow-up phase will commence for all subjects that achieve complete wound closure, which is designed to measure longevity and durability of the closed wound. This follow-up period will consist of a four-week follow-up with two visits at each two-week interval.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form.
2. Male or female patient at least 18 years of age or older, as of the date of the screening visit.
3. Has a VLU between the knee and ankle (at or above the malleoli), with a surface area in the range of ≥ 2.0 cm2 and ≤ 20.0 cm2 when measured by the investigator staff at the screening visit using the eKare device post debridement.

   1. If the subject presents with > 1, but ≤ 3 VLU on the same leg, the largest ulcer will be selected as the target ulcer.
   2. If the target ulcer is < 1cm from another VLU, the ulcers should be traced as a single target ulcer provided at least one of the ulcers is at least 2.0 cm2 in area and the total surface area of the VLUs is ≤ 20.0 cm2.
4. Target ulcer involves a full-thickness skin loss, but without exposure of tendon, muscle, or bone.
5. Target ulcer duration ≥ 4 weeks but ≤ 52 weeks (12 months).
6. Venous insufficiency confirmed by duplex Doppler ultrasound examining valvular or venous incompetence.

   a. Availability of a complete report of a previous examination performed 12 months of screening will be acceptable, and this examination would not be required to be repeated.
7. Arterial supply adequacy confirmed by any one of the following:

   1. Great toe pressure ≥ 50 mm/Hg
   2. Systolic blood pressure Ankle Brachial Index (ABI) in the range ≥ 0.80 ≤ 1.10
   3. TcPO2 ≥ 40 mmHg from the foot
8. Willing to follow all instructions given by the Investigator, return for all visits, and adhere to compression protocols while on the study.

Exclusion Criteria:

1. A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
2. Acute Deep Vein Thrombosis (DVT), defined as the first 10 days from onset of symptoms, or any DVT for which compression is considered by the Investigator to be contraindicated.
3. Clinical evidence of ulcer bed infection, or infected hardware.
4. Documented history of osteomyelitis at the target ulcer location within six (6) months preceding the screening visit.
5. Refusal or inability to tolerate compression therapy.
6. Pregnant women.
7. Women of child-bearing potential who are unwilling to avoid pregnancy or use an effective form of birth control.
8. Hemoglobin A1c (HbA1c) level is > 12% (108 mmol/mol).
9. Current therapy with systemic antibiotics.
10. Current therapy with cytotoxic agents.
11. Current therapy with chronic (> 10 days) oral corticosteroids.
12. Current therapy with TNFα inhibitors other than Trental® (pentoxifylline).
13. Has tested positive for Human Immunodeficiency Virus (HIV) or has Acquired Immune Deficiency Syndrome (AIDS).
14. Has malignancy or history of cancer in the preceding 5 years other than non-melanoma skin cancer.
15. Currently on dialysis or planning to start dialysis.
16. Is currently enrolled or participated in another device, drug, or biological trial within 30 days of screening.
17. Therapy of the target ulcer with other birth tissue products, autologous skin graft, Apligraf®, or Dermagraft® within 30 days preceding the screening visit.
18. Therapy of the target ulcer with topical growth factors within thirty (30) days preceding the screening visit.
19. Any previous use of Vendaje®, Vendaje AC®, AmnioWrap2® applied to the target ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To determine whether non-ischemic, non-infected VLUs treated with standard care plus BR-AC results in a higher probability of achieving complete wound closure compared to standard care alone. | over the 12-week treatment period
  Percentage of subjects with complete wound closure over the 12-week treatment period, defined as 100% reepithelialization

SECONDARY OUTCOMES:
To compare differences between treatment groups in proportions of wounds with complete wound closure, based on time in days to closure | at 12 weeks
  Percent change from baseline in wound surface area (cm2) at 12-weeks post-randomization
To compare differences between treatment groups in percent change in wound area (cm2) | at 12 weeks
  Percent change from baseline in wound surface area (cm2) at 12-weeks post-randomization
To determine the total number of applications of BR-AC needed to achieve complete wound closure | at 12 weeks
  Percent change from baseline in wound volume (cm3) at 12-weeks post-randomization
To determine whether subjects that crossover and receive standard care plus BR-AC results in a higher probability of achieving complete wound closure over the 12 additional weeks versus standard care alone | over an additional 12 weeks
  Time in days from Visit 18 to initial observation of wound closure (defined as 100% reepithelialization of the wound without drainage) over an additional 12 weeks (Visits 19-30), where healing has been confirmed at two visits two weeks apart

OTHER OUTCOMES:
Number of participants that acquire clinical signs and symptoms of infections post-randomization | over 12-weeks post-randomization
  Differences in clinical signs and symptoms of infection from Visit 2 through end of study between the treatment groups
Proportion of subjects experiencing adverse events, by treatment group | over the 17-week study period
  Spontaneously reported and elicited adverse events, coded in MedDRA

CONTACTS AND LOCATIONS:
Overall Officials: Bert Slade, MD, Study Director — Independent
Locations (23):
- United States (23):
  - Site 17, Guntersville, Alabama
  - Site 2b, Castro Valley, California
  - Site 19b, Glendale, California
  - Site 36, Oxnard, California
  - Site 37, Oxnard, California
  - Site 19, Palmdale, California
  - Site 02, San Francisco, California
  - Site 2a, San Francisco, California
  - Site 04, Sylmar, California
  - Site 30, Torrance, California
  - Site 01, Vista, California
  - Site 34, Aventura, Florida
  - Site 27, Coral Gables, Florida
  - Site 20, Deerfield Beach, Florida
  - Site 33, Fort Walton Beach, Florida
  - Site 35, Miami, Florida
  - Site 31, Miami, Florida
  - Site 06, O'Fallon, Illinois
  - Site 18, Boston, Massachusetts
  - Site 32, St Louis, Missouri
  - Site 16, Lake Success, New York
  - Site 38, Corpus Christi, Texas
  - Site 03, Fort Worth, Texas